CLINICAL TRIAL: NCT01083069
Title: Neurological Outcome After Mild Induced Hypothermia (MIH) After Restoration of Spontaneous Circulation
Brief Title: Follow up After Survived Therapy With Mild Induced Hypothermia (MIH) After Restoration of Spontaneous Circulation (ROSC)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Leipzig (Other)
Responsible Party: Holger Thiele, Associate Professor Study Chair, University of Leipzig, Heart center
Other Study IDs: Cool-Trial Follow up
Record Dates: First submitted 2010-02-25; First posted 2010-03-09 (Estimated); Last update posted 2010-03-09 (Estimated); Status verified 2010-01

CONDITIONS: Cardiac Arrest; Hypothermia
Keywords: Sudden cardiac arrest; hypothermia; neurological outcome
MeSH Terms: conditions — Heart Arrest; Hypothermia; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COOL: Patients after therapy with mild hypothermia
- UnCool: Patients without therapy with mild hypothermia due to non-operational cooling-devices

SUMMARY:
Sudden cardiac arrest (SCA) remains one of the major leading causes of death. Cognitive deficits are common in survivors of SCA. Postresuscitative mild induced hypothermia (MIH) lowers mortality and reduces neurologic damage after cardiac arrest. The investigators evaluated the long term neurological outcome after mild hypothermia after restoration of spontaneous circulation.

DETAILED DESCRIPTION:
Consecutive patients with restoration of spontaneous circulation (ROSC) after resuscitation due to out-of-hospital SCA, admitted to our intensive care unit, underwent MIH. Hypothermia was induced by infusion of cold saline and whole-body-cooling methods (electronic randomization: invasive Coolgard or non-invasive ArcticSun). The core body temperature was operated at 32 to 34 °C over a period of 24 hours followed by active rewarming. Neurological status was evaluated at hospital discharge and 6 months after discharge using the Pittsburgh Cerebral Performance Category (CPC).

ELIGIBILITY:
Inclusion Criteria:

* survived cardiac arrest
* voluntary consent

Exclusion Criteria:

* no voluntary consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients after restoration of spontaneous circulation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Neurological outcome after 6 month after MIH, Quality of life-survey | 6 Month
  Neurological outcome after 6 month after MIH measured by questionnaire.

SECONDARY OUTCOMES:
Managing daily activities | 6 Month
  Managing daily activities after 6 month after tMIH measured with a questionnaire.
Surviving after hospitalization | 6 Month
  Surviving after hospitalization after MIH
Neurological outcome depending of the beginning of MIH | 6 month
  Neurological outcome depending of the beginning of MIH
Neurological Outcome in consideration of the practice of the treating instances. | 6 month
  Neurological outcome in consideration of the practice of the treating instances after restoration of spontanous circulation measured with a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Holger Thiele, Associate Professor, Principal Investigator — Study Chair; Undine Pittl, MD, Study Director — Study Sub-invesigator
Locations (1):
- University of Leipzig, Heart Center, Cardiology, Leipzig, Germany